CLINICAL TRIAL: NCT01839487
Title: A Phase 2, Randomized, Multicenter Study of PEGPH20 (PEGylated Recombinant Human Hyaluronidase) Combined With Nab-Paclitaxel Plus Gemcitabine Compared With Nab-Paclitaxel Plus Gemcitabine in Subjects With Stage IV Previously Untreated Pancreatic Cancer
Brief Title: PEGPH20 Plus Nab-Paclitaxel Plus Gemcitabine Compared With Nab-Paclitaxel Plus Gemcitabine in Participants With Stage IV Untreated Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HALO-109-202
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Results first posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: pancreatic ductal carcinoma(PDA); Pancreatic ductal carcinoma; PEGPH20; Gemcitabine; Nab-paclitaxel
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Pancreatic Ductal | interventions — PEGPH20; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Dexamethasone; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Run-in Phase - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine (Experimental): Participants will receive 3.0 micrograms/kilogram (mcg/kg) PEGPH20 with 125 milligrams/square meter (mg/m^2) NAB and 1000 mg/m^2 GEM as intravenous (IV) infusion. In Cycle 1 Week 1, PEGPH20 will be administered alone on Days 1 and 4 and NAB+GEM will be given on Day 2 at approximately 24 hours after first dose of PEGPH20. In Cycle 1 Weeks 2 and 3, PEGPH20 will be given twice/week on Days 8, 11, 15 and 18 and NAB+GEM will be given once/week at 2 to 4 hours after PEGPH20 administration on Days 8 and15. In Cycle 2 onwards, PEGPH20, NAB, and GEM will be given once/week on Days 1 8 and 15. NAB+GEM will be given 2 to 4 hours after PEGPH20 dose. Each cycle will be of 4-weeks with Week 4 of every cycle as a rest week (no treatment will be given). Treatment will continue until documented disease progression or unacceptable toxicity. Dexamethasone 8 mg will be given in each cycle within 2 hours prior and 8 to 12 hours after completion of each PEGPH20 infusion.
  Interventions: Drug: PEGPH20; Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Dexamethasone
- Run-in Phase - AG: Nab-paclitaxel + Gemcitabine (Active Comparator): Participants will receive 125 mg/m^2 NAB and 1000 mg/m^2 GEM, as an IV infusion once weekly on Days 1, 8, and 15 of each cycle. Each cycle will be of 4-weeks (28 days) with Week 4 of every cycle as a rest week (that is; no treatment will be given). Treatment will continue until documented disease progression or unacceptable toxicity. Dexamethasone 8 mg will be given in each cycle within 2 hours prior to the beginning of each NAB infusion and 8 to 12 hours after the completion of GEM infusion.
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Dexamethasone
- Phase 2: Stage 1 - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine (Experimental): Participants will receive 3.0 mcg/kg PEGPH20 with 125 mg/m^2 NAB and 1000 mg/m^2 GEM as an IV infusion. In Cycle 1 Week 1, PEGPH20 will be given alone on Days 1 and Day 4 and NAB+GEM will be given on Day 2 at approximately 24 hours after first dose of PEGPH20. In Cycle 1 Weeks 2 and 3, PEGPH20 will be given twice/week on Days 8, 11, 15, and 18 and NAB+GEM will be given once/week at 2 to 4 hours after PEGPH20 administration on Days 8 and 15. In Cycle 2 onwards, PEGPH20, NAB, and GEM will be given once/week on Days 1, 8, and 15. NAB+GEM will be given 2 to 4 hours after dose of PEGPH20. Each cycle will be of 4-weeks with Week 4 of every cycle as a rest week (no treatment will be given). Treatment will continue until documented disease progression or unacceptable toxicity. Dexamethasone 8 mg will be given in each cycle within 2 hours prior to the beginning and 8 to 12 hours after the completion of each PEGPH20 infusion.
  Interventions: Drug: PEGPH20; Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Dexamethasone
- Phase 2: Stage 1 - AG: Nab-paclitaxel + Gemcitabine (Active Comparator): Participants will receive 125 mg/m^2 NAB and 1000 mg/m^2 GEM as an IV infusion once weekly on Days 1, 8, and 15 of each cycle. Each cycle will be of 4-weeks (28 days) with Week 4 of every cycle as a rest week (that is; no treatment will be given). Treatment will continue until documented disease progression or unacceptable toxicity. Dexamethasone 8 mg will be given in each cycle within 2 hours prior to the beginning of each NAB infusion and 8 to 12 hours after the completion of GEM infusion.
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Dexamethasone
- Phase 2: Stage 2 - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine (Experimental): Participants will receive 3.0 mcg/kg PEGPH20 with 125 mg/m^2 NAB and 1000 mg/m^2 GEM as an IV infusion. In Cycle 1 Week 1, PEGPH20 will be given alone on Days 1 and 4 and NAB+GEM will be given on Day 2 at approximately 24 hours after first dose of PEGPH20. In Cycle 1 Weeks 2 and 3, PEGPH20 will be given twice/week on Days 8, 11, 15, and 18 and NAB+GEM will be given once/week at 2 to 4 hours after PEGPH20 administration on Days 8 and 15. In Cycle 2 onwards, PEGPH20, NAB, and GEM will be given once/week on Days 1, 8, and 15. NAB+GEM will be given 2 to 4 hours after dose of PEGPH20. Each cycle will be of 4-weeks with Week 4 of every cycle as a rest week (no treatment will be given). Treatment will continue until documented disease progression or unacceptable toxicity. Dexamethasone 8 mg will be given in each cycle within 2 hours prior to beginning and 8 to 12 hours after completion of each PEGPH20 infusion. Enoxaparin 40 mg/day or 1 mg/kg/day will be given subcutaneously (SC).
  Interventions: Drug: PEGPH20; Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Dexamethasone; Drug: Enoxaparin
- Phase 2: Stage 2 - AG: Nab-paclitaxel + Gemcitabine (Active Comparator): Participants will receive 125 mg/m^2 NAB and 1000 mg/m^2 GEM as an IV infusion once weekly on Days 1, 8, and 15 of each cycle. Each cycle will be of 4-weeks (28 days) with Week 4 of every cycle as a rest week (that is; no treatment will be given). Treatment will continue until documented disease progression or unacceptable toxicity. Dexamethasone 8 mg will be given in each cycle within 2 hours prior to the beginning of each NAB infusion and 8 to 12 hours after the completion of GEM infusion. Enoxaparin 40 mg/day or 1 mg/kg/day will be given SC.
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Dexamethasone; Drug: Enoxaparin

INTERVENTIONS:
Drug: PEGPH20 — PEGPH20 will be administered as per the dose and schedule specified in the respective arms.
  Arms: Phase 2: Stage 1 - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine; Phase 2: Stage 2 - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine; Run-in Phase - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine
Drug: Nab-paclitaxel — Nab-paclitaxel will be administered as per the dose and schedule specified in the respective arms.
  Other Names: Abraxane
Drug: Gemcitabine — Gemcitabine will be administered as per the dose and schedule specified in the respective arms.
  Other Names: Gemzar
Drug: Dexamethasone — Dexamethasone will be administered as per the dose and schedule specified in the respective arms.
Drug: Enoxaparin — Enoxaparin will be administered as per the dose and schedule specified in the respective arms.
  Arms: Phase 2: Stage 2 - AG: Nab-paclitaxel + Gemcitabine; Phase 2: Stage 2 - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine

SUMMARY:
This study is designed to compare the treatment effect of PEGPH20 combined with nab-paclitaxel (NAB) and gemcitabine (GEM) [PAG] to NAB and GEM [AG] in participants with Stage IV previously untreated pancreatic ductal adenocarcinoma (PDA).

The study will have 2 run-in phases, one for each formulation of PEGPH20 (original and new formulations), and a Phase 2 portion. The 2 run-in phases will evaluate the safety and tolerability of the PAG treatment using the original and new succinic acid PEGPH20 formulation, respectively, compared with AG treatment. Phase 2 will have 2 stages due to a partial clinical hold that occurred from April through July 2014. The participants will be randomized in 3:1 for the run-in phases. The first stage will randomize participants in a 1:1 ratio. The second stage will randomize participants in a 2:1 ratio (PAG:AG).

This is an open-label study. To minimize bias to the progression-free survival endpoint, disease progression will be based on the assessment of the Central Imaging Reader (CIR). Determination of clinical progression by the Investigator without corresponding CIR confirmation will be documented with the relevant signs and symptoms.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed Informed consent.
* Histologically confirmed Stage IV PDA with documented disseminated neoplasm to liver and /or lung. Must have archival or fresh tissue (block /slides) available pre-dose.
* One or more metastatic tumors measurable on computed tomography (CT) scan per RECIST v.1.1 , excluding the primary pancreatic lesion.
* No previous radiotherapy, surgery, chemotherapy or investigational therapy for the treatment of metastatic disease.
* Karnofsky Performance Status greater than or equal to (≥) 70%.
* Life expectancy ≥3 months.
* Age ≥18 years.
* Screening laboratory values of hemoglobin, platelets, absolute neutrophil count (ANC), bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), serum creatinine, serum albumin, prothrombin time/international normalized ratio (INR), and partial thromboplastin time (PTT) within specified values/criteria per protocol prior to dosing.

Key Exclusion Criteria:

* Non-metastatic PDA.
* Evidence of deep vein thrombosis (DVT), pulmonary embolism (PE), or other known thromboembolic event present during screening period.
* Known central nervous system involvement or brain metastasis.
* New York (NY) Heart Association Class III or IV cardiac disease or myocardial infarction within the past 12 months.
* Prior history of cerebrovascular accident or transient ischemic attack.
* Pre-existing carotid artery disease.
* Active, uncontrolled bacterial, viral, or fungal infection requiring systemic therapy.
* Current use of megestrol acetate (use within 10 days of Day 1).
* Known infection with human immunodeficiency virus, Hepatitis B, or Hepatitis C.
* History of another primary cancer within the last 3 years with the exception of non-melanoma skin cancer, early state prostate cancer, or curatively-treated cervical cancer in-situ.
* Contraindication to heparin as per National Comprehensive Cancer Network (NCCN) guidelines.
* Previous major bleed (bleeding requiring transfusion of red blood cells) on low-molecular weight heparin (LMWH).
* Any other disease, metabolic dysfunction, physical examination finding or clinical laboratory finding that leads to reasonable suspicion of disease or condition that contraindicates the use of an investigational drug, that may affect interpretation of results, or render the participant at a high risk of treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2013-05-14 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP, Clinical Development, Study Director — Halozyme Therapeutics
Locations (51):
- United States (51):
  - Alabama Oncology, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - Arizona Oncology Associates, PC, Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Providence St Joseph Medical Center, Burbank, California
  - Scripps Cancer Center, La Jolla, California
  - UCSD - Moore's Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Medical Center, Orange, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Stamford Hospital, Stamford, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Miami, Sylvester comprehensive Cancer Center, Miami, Florida
  - H. Lee Moffit Cancer Center, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Norton Cancer Institute - Norton HealthCare Pavilion, Louisville, Kentucky
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Mass Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Unniversity of Minnesota, Minneapolis, Minnesota
  - Research Medical Center, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore Long Island Jewish Health System, Lake Success, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Gabrail Cancer Center, Canton, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Texas Oncology - Baylor, Dallas, Texas
  - Cancer Care Centers of South Texas, New Braunfels, Texas
  - Texas Oncology, Tyler, Texas
  - Columbia Basin Hematology and Oncology, Kennewick, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - NorthWest Medical Specialties, PLLC, Tacoma, Washington
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin
  - Froedtert Hospital, Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Hingorani SR, Zheng L, Bullock AJ, Seery TE, Harris WP, Sigal DS, Braiteh F, Ritch PS, Zalupski MM, Bahary N, Oberstein PE, Wang-Gillam A, Wu W, Chondros D, Jiang P, Khelifa S, Pu J, Aldrich C, Hendifar AE. HALO 202: Randomized Phase II Study of PEGPH20 Plus Nab-Paclitaxel/Gemcitabine Versus Nab-Paclitaxel/Gemcitabine in Patients With Untreated, Metastatic Pancreatic Ductal Adenocarcinoma. J Clin Oncol. 2018 Feb 1;36(4):359-366. doi: 10.1200/JCO.2017.74.9564. Epub 2017 Dec 12. PMID 29232172
- [Derived] Wang S, Bager CL, Karsdal MA, Chondros D, Taverna D, Willumsen N. Blood-based extracellular matrix biomarkers as predictors of survival in patients with metastatic pancreatic ductal adenocarcinoma receiving pegvorhyaluronidase alfa. J Transl Med. 2021 Jan 21;19(1):39. doi: 10.1186/s12967-021-02701-z. PMID 33478521
- See also: Reflects interim analysis conducted on mature data when 95% of participants had discontinued from the study. — https://pubmed.ncbi.nlm.nih.gov/29232172/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study had 2 run-in phases (for evaluating safety and tolerability of PAG [PEGPH20 + Nab-paclitaxel {NAB} + Gemcitabine {GEM}] treatment), one for each formulation of PEGPH20 (original and new formulations [injectable solution containing 3.5 milligrams/milliliter {mg/mL} and 0.3 mg/mL PEGPH20, respectively]), and a Phase 2 (Stage 1 and 2) portion.
Pre-assignment Details: Study was on partial clinical hold from April to July 2014 due to higher incidence of thromboembolic events (TE) in PAG arm participants. Study enrollment (Stage 2) was reopened in June 2014 after excluding participants with high-risk of TE and adding enoxanparin prophylasis. Participants of PAG and AG arm both received AG during clinical hold.
Groups:
- Run-in Phase - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine: Participants received 3.0 micrograms/kilogram (mcg/kg) PEGPH20 with 125 milligrams/square meter (mg/m^2) nab-paclitaxel (NAB) and 1000 mg/m^2 gemcitabine (GEM) as intravenous (IV) infusion. In Cycle 1 Week 1, PEGPH20 was given alone on Days 1 and 4 and NAB+GEM was given on Day 2 at approximately 24 hours after first dose of PEGPH20. In Cycle 1 Weeks 2 and 3, PEGPH20 was given twice/week on Days 8, 11, 15, 18 and NAB+GEM were given once/week at 2 to 4 hours after PEGPH20 administration on Days 8 and 15. In Cycle 2 onwards, PEGPH20, NAB, and GEM were given once/week on Days 1, 8, and 15. NAB+GEM were given 2 to 4 hours after PEGPH20 dose. Each cycle was of 4-weeks with Week 4 of every cycle as a rest week (no treatment was given). Treatment was continued until documented disease progression or unacceptable toxicity. Dexamethasone 8 mg was given in each cycle within 2 hours prior to beginning and 8 to 12 hours after completion of each PEGPH20 infusion.
- Run-in Phase - AG: Nab-paclitaxel + Gemcitabine; Phase 2: Stage 1 - AG: Nab-paclitaxel + Gemcitabine: Participants received 125 mg/m^2 NAB and 1000 mg/m^2 GEM as an IV infusion once weekly on Days 1, 8, and 15 of each cycle. Each cycle was of 4-weeks (28 days) with Week 4 of every cycle as a rest week (that is; no treatment was given). Treatment was continued until documented disease progression or unacceptable toxicity. Dexamethasone 8 mg was given in each cycle within 2 hours prior to the beginning of each NAB infusion and 8 to 12 hours after the completion of GEM infusion.
- Phase 2: Stage 1 - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine: Participants received 3.0 mcg/kg PEGPH20 with 125 mg/m^2 NAB and 1000 mg/m^2 GEM as an IV infusion. In Cycle 1 Week 1, PEGPH20 was given alone on Days 1 and 4 and NAB+GEM was given on Day 2 at approximately 24 hours after the first dose of PEGPH20. In Cycle 1 Weeks 2 and 3, PEGPH20 was given twice/week on Days 8, 11, 15, and 18 and NAB+GEM were given once/week at 2 to 4 hours after PEGPH20 administration on Days 8 and 15. In Cycle 2 onwards, PEGPH20, NAB, and GEM were administered once/week on Days 1, 8, and 15. NAB+GEM were given 2 to 4 hours after the dose of PEGPH20. Each cycle was of 4-weeks (28 days) with Week 4 of every cycle as a rest week (that is; no treatment was given). Treatment was continued until documented disease progression or unacceptable toxicity. Dexamethasone 8 mg was given in each cycle within 2 hours prior to the beginning and 8 to 12 hours after the completion of each PEGPH20 infusion.
- Phase 2: Stage 2 - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine: Participants received 3.0 mcg/kg PEGPH20 with 125 mg/m^2 NAB and 1000 mg/m^2 GEM as an IV infusion. In Cycle 1 Week 1, PEGPH20 was given alone on Days 1 and 4 and NAB+GEM was given on Day 2 at approximately 24 hours after the first dose of PEGPH20. In Cycle 1 Weeks 2 and 3, PEGPH20 was given twice/week on Days 8, 11, 15, and 18 and NAB+GEM were given once/week at 2 to 4 hours after PEGPH20 administration on Days 8 and 15. In Cycle 2 onwards, PEGPH20, NAB, and GEM were given once/week on Days 1, 8, and 15. NAB+GEM were given 2 to 4 hours after dose of PEGPH20. Each cycle was of 4-weeks with Week 4 of every cycle as a rest week (no treatment was given). Treatment was continued until documented disease progression or unacceptable toxicity. Dexamethasone 8 mg was given in each cycle within 2 hours prior to beginning and 8 to 12 hours after completion of each PEGPH20 infusion. Enoxaparin 40 mg/day or 1 mg/kg/day was given subcutaneously (SC).
- Phase 2: Stage 2 - AG: Nab-paclitaxel + Gemcitabine: Participants received 125 mg/m^2 NAB and 1000 mg/m^2 GEM as an IV infusion once weekly on Days 1, 8, and 15 of each cycle. Each cycle was of 4-weeks (28 days) with Week 4 of every cycle as a rest week (that is; no treatment was given). Treatment was continued until documented disease progression or unacceptable toxicity. Dexamethasone 8 mg was given in each cycle within 2 hours prior to the beginning of each NAB infusion and 8 to 12 hours after the completion of GEM infusion. Enoxaparin 40 mg/day or 1 mg/kg/day was given SC.
Period: Run-in Phase (Maximum Exposure:295 Days)
Arm/Group | Run-in Phase - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine | Run-in Phase - AG: Nab-paclitaxel + Gemcitabine | Phase 2: Stage 1 - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine | Phase 2: Stage 1 - AG: Nab-paclitaxel + Gemcitabine | Phase 2: Stage 2 - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine | Phase 2: Stage 2 - AG: Nab-paclitaxel + Gemcitabine
Started | 16 | 7 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 16 | 7 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 14 | 6 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other than specified | 1 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 (Maximum Exposure:935 Days)
Arm/Group | Run-in Phase - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine | Run-in Phase - AG: Nab-paclitaxel + Gemcitabine | Phase 2: Stage 1 - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine | Phase 2: Stage 1 - AG: Nab-paclitaxel + Gemcitabine | Phase 2: Stage 2 - PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine | Phase 2: Stage 2 - AG: Nab-paclitaxel + Gemcitabine
Started | 0 | 0 | 61 | 62 | 89 | 44
Completed | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 61 | 62 | 88 | 44
Not completed — Withdrawal by Subject | 0 | 0 | 12 | 9 | 4 | 8
Not completed — Death | 0 | 0 | 46 | 49 | 71 | 32
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 1 | 10 | 3
Not completed — Other than specified | 0 | 0 | 1 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized, including the run-in phases.
Groups:
- PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine: Participants received 3.0 mcg/kg PEGPH20 with 125 mg/m^2 NAB and 1000 mg/m^2 GEM as an IV infusion. In Cycle 1 Week 1, PEGPH20 was given alone on Days 1 and 4 and NAB+GEM was given on Day 2 at approximately 24 hours after the first dose of PEGPH20. In Cycle 1 Weeks 2 and 3, PEGPH20 was given twice/week on Days 8, 11, 15, and 18 and NAB+GEM were given once/week at 2 to 4 hours after PEGPH20 administration on Days 8 and 15. In Cycle 2 onwards, PEGPH20, NAB, and GEM were given once/week on Days 1, 8, and 15. NAB+GEM were given 2 to 4 hours after the dose of PEGPH20. Each cycle was of 4-weeks (28 days) with Week 4 of every cycle as a rest week (that is; no treatment was given). Treatment was continued until documented disease progression or unacceptable toxicity. Dexamethasone 8 mg was given in each cycle within 2 hours prior to the beginning and 8 to 12 hours after the completion of each PEGPH20 infusion.
- AG: Nab-paclitaxel + Gemcitabine: Participants received 125 mg/m^2 NAB and 1000 mg/m^2 GEM as an IV infusion once weekly on Days 1, 8, and 15 of each cycle. Each cycle was of 4-weeks (28 days) with Week 4 of every cycle as a rest week (that is; no treatment was given). Treatment was continued until documented disease progression or unacceptable toxicity. Dexamethasone 8 mg was given in each cycle within 2 hours prior to the beginning of each NAB infusion and 8 to 12 hours after the completion of GEM infusion.
- Total: Total of all reporting groups
Arm/Group | PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine | AG: Nab-paclitaxel + Gemcitabine | Total
Number analyzed (Participants) | 166 | 113 | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (9.72) | 65.0 (8.82) | 64.6 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 58 | 123
  Male | 101 | 55 | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 13
  Not Hispanic or Latino | 160 | 104 | 264
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 11 | 9 | 20
  White | 146 | 91 | 237
  More than one race | 1 | 7 | 8
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS: time from randomization until first occurrence of disease progression, either by central radiologic determination (Response Evaluation Criteria in Solid Tumours [RECIST] version 1.1) or by clinical progression determined by Investigator, or death during treatment period from any cause. Radiological disease progression was defined as at least a 20 percent (%) increase in sum of diameters of target lesions, taking as reference the smallest sum on study thus far, nadir (this included baseline sum if that was the smallest on study); Sum must also demonstrate an absolute increase of at least 5 millimeters (mm); Appearance of one or more new lesions; Unequivocal progression of existing non-target lesions. Surviving participants without disease progression were censored for PFS analysis at the date of last evaluable post-baseline tumor assessment. Surviving participants without any post-baseline disease assessment were censored on Day 1. PFS was estimated using Kaplan-Meier (KM) method.
Time Frame: From the date of randomization until disease progression or death from any cause (maximum exposure: 30.72 months for PAG, and 20.27 months for AG)
Population: Efficacy evaluable (EE) population: all randomized participants who received at least 1 dose of any study drug, who had measurable disease at baseline, and had a post-baseline response assessment, or had clinical disease progression without a post-baseline computed tomography (CT) scan, or had died on or prior to 14 days after the last dose date.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine | AG: Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 139 | 92
months | 6.05 [5.36 to 7.20] | 5.26 [3.91 to 6.54]
Statistical Analysis 1: Comparison: PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine vs AG: Nab-paclitaxel + Gemcitabine; Hazard ratio PAG/AG was based on Cox proportional hazards model stratified by the Karnofsky Performance Status (KPS) category (70-80% and 90-100%) at screening using AG as the reference arm; Test type: Other; p = 0.058, Log Rank — Threshold for significance at 0.1 level; P-value was based on stratified log-rank test with the KPS category at screening as the stratification factor; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.54 to 1.01]

2. Primary Outcome: Percentage of Participants in the PAG Arm Who Experienced Any Thromboembolic (TE) Event in Stage 2 of the Study
Description: TE events were identified by applying the Medical Dictionary for Regulatory Activities (MedDRA) Standardized MedDRA Queries (SMQ) search strategy for 3 SMQs: TE arterial, TE venous, and TE vessel type unspecified and mixed arterial and venous. TE events were considered by the Sponsor to be adverse events (AEs) of special interest. All TE events, regardless of type of event, severity, or seriousness were reported. Participants with multiple events were counted only once. A summary of serious and all other non-serious adverse events regardless of causality is located in the 'Reported AE section'.
Time Frame: From first exposure to any study drug (PEGPH20, NAB, GEM) through 30 days after end of treatment visit (maximum exposure: 30.72 months for PAG)
Population: Safety population of Stage 2 included all participants enrolled in Stage 2 of Phase 2 of study after the clinical hold, and who received at least 1 dose of study drug. This outcome was planned to be reported only for PAG arm as pre-specified in protocol.
Measure: Number; unit: percentage of participants
Arm/Group | PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 86
percentage of participants | 14.0

3. Secondary Outcome: PFS in Relation to Tumor Hyaluronan (HA) Levels
Description: PFS was defined as time from randomization until first occurrence of disease progression, either by central radiologic determination (RECIST version 1.1) or by clinical progression determined by Investigator, or death during treatment period from any cause. Disease progression was defined as at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study thus far, nadir (this included baseline sum if that was the smallest on study); Sum must also demonstrate an absolute increase of at least 5 mm; Appearance of one or more new lesions; Unequivocal progression of existing non-target lesions. Surviving participants without disease progression were censored for PFS analysis at the date of last evaluable post-baseline tumor assessment. Surviving participants without any post-baseline disease assessment were censored on Day 1. PFS was estimated using KM method. PFS was measured in HA-high and HA-low participants.
Time Frame: as for outcome 1
Population: Intent-to -treat (ITT) population included all participants who were randomized, including the run-in phases. 'Number analyzed'=participants with HA-high or HA-low levels.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine | AG: Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 153 | 93
months
  HA-High: number analyzed (Participants) | 49 | 35
  HA-High | 9.23 [5.98 to 10.55] | 5.19 [3.52 to 6.54]
  HA-Low: number analyzed (Participants) | 104 | 58
  HA-Low | 5.59 [4.70 to 7.03] | 5.26 [3.78 to 7.33]
Statistical Analysis 1: Comparison: PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine vs AG: Nab-paclitaxel + Gemcitabine; Hazard ratio PAG/AG for HA-high was based on Cox proportional hazards model stratified by the KPS category (70-80% and 90-100%) at screening using AG as the reference arm; Test type: Other; p = 0.092, Log Rank — Threshold for significance at 0.1 level; P-value was based on stratified log-rank test with the KPS category at screening as the stratification factor; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.30 to 1.10]
Statistical Analysis 2: Comparison: PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine vs AG: Nab-paclitaxel + Gemcitabine; Hazard ratio PAG/AG for HA-low was based on Cox proportional hazards model stratified by the KPS category (70-80% and 90-100%) at screening using AG as the reference arm; Test type: Other; p = 0.514, Log Rank — Threshold for significance at 0.1 level; P-value was based on stratified log-rank test with the KPS category at screening as the stratification factor; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.59 to 1.31]

4. Secondary Outcome: Objective Response Rate (ORR): Percentage of Participants With Objective Response
Description: ORR was defined as percentage of participants who achieved either a complete response (CR) or partial response (PR) regardless of confirmation, as assessed by RECIST version 1.1. CR was defined as disappearance of all target and non-target lesions; Any pathological or non-pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of randomization until last date on study treatment (maximum exposure: 30.72 months for PAG, and 20.27 months for AG)
Population: ITT population included all participants who were randomized, including the run-in phases.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine | AG: Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 166 | 113
percentage of participants | 40.4 [32.83 to 48.24] | 32.7 [24.21 to 42.21]
Statistical Analysis 1: Comparison: PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine vs AG: Nab-paclitaxel + Gemcitabine; p-Value and relative risk were based on a stratified Cochran-Mantel-Haenszel method using KPS category at screening as the stratification factor; Test type: Other; p = 0.225, Cochran-Mantel-Haenszel — Threshold for significance at 0.1 level; Risk Ratio (RR) = 1.22, 95% CI 2-sided [0.88 to 1.68]

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization until death from any cause. Participants who died or were lost to follow-up by the date of analysis data cutoff were censored at their last contact date.
Time Frame: From randomization until death from any cause (maximum exposure: 30.72 months for PAG, and 20.27 months for AG)
Population: ITT population included all participants who were randomized, including the run-in phases.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine | AG: Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 166 | 113
months | 9.59 [8.15 to 12.06] | 9.23 [7.59 to 10.71]
Statistical Analysis 1: Comparison: PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine vs AG: Nab-paclitaxel + Gemcitabine; Hazard ratio PAG/AG was based on Cox proportional hazards model stratified by the KPS category (70-80% and 90-100%) at screening using AG as the reference arm; Test type: Other; p = 0.495, Log Rank — Threshold for significance at 0.1 level; P-value was based on stratified log-rank test with the KPS category at screening as the stratification factor; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.70 to 1.19]

6. Secondary Outcome: Percentage of Participants With AEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: From first exposure to any study drug (PEGPH20, NAB, GEM) through 30 days after end of treatment visit (maximum exposure: 30.72 months for PAG and 20.27 months for AG)
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine | AG: Nab-paclitaxel + Gemcitabine
Number analyzed (Participants) | 160 | 100
percentage of participants | 99.4 | 98.0

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PEGPH20
Description: Samples were analyzed for PEGPH20 concentration using a validated electrochemiluminescence immunoassay. Plasma samples to assess the potential effects of NAB+GEM on PEGH20 pharmacokinetic (PK) were collected in the PAG treatment group in the run-in phases (Run-in Phase 1: Original PEGPH20 formulation [3.5 mg/mL], and Run-in Phase 2: New PEGPH20 formulation [0.3 mg/mL]).
Time Frame: Pre-PEGPH20 dosing and 15 minutes, 1 hour, 2 hours, and 4 hours post-PEGPH20 dosing on Days 1 and 15 of Cycle 1
Population: PK analysis population included all participants who received any part of a dose of PEGPH20 and had measurable PEGPH20 concentrations in at least 1 sample collected for PK analysis. 'Number analyzed'=participants evaluable for this outcome at specified timepoints.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Groups:
- Run-in Phase 1-PAG: PEGPH20 (Original Formulation) + NAB + GEM; Run-in Phase 2- PAG: PEGPH20 (New Formulation) + NAB + GEM: Participants received 3.0 mcg/kg PEGPH20 with 125 mg/m^2 NAB, and 1000 mg/m^2 GEM, as IV infusion. In Cycle 1 Week 1, PEGPH20 was administered alone on Day 1, 4, and NAB+GEM were administered on Day 2, approximately 24 hours after first dose of PEGPH20. In Cycle 1 Weeks 2 and 3, PEGPH20 was given twice/week on Days 8, 11, 15, 18, and NAB+GEM were given once/week, 2 to 4 hours after PEGPH20 administration on Days 8, 15. In Cycle 2 onwards, PEGPH20, NAB, and GEM were given once/week on Days 1, 8, 15. NAB+GEM were given 2 to 4 hours after PEGPH20 dose. Each treatment cycle was of 4-weeks with Week 4 of every cycle as a rest week (no treatment). Treatment was continued until disease progression or unacceptable toxicity. Dexamethasone 8 mg was administered in each treatment cycle within 2 hours prior to beginning of each PEGPH20 infusion and 8 to 12 hours after completion of each PEGPH20 infusion.
Arm/Group | Run-in Phase 1-PAG: PEGPH20 (Original Formulation) + NAB + GEM | Run-in Phase 2- PAG: PEGPH20 (New Formulation) + NAB + GEM
Number analyzed (Participants) | 6 | 8
nanograms/milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 5 | 8
  Day 1 | 72.1 (16.90) | 67.8 (17.60)
  Day 15: number analyzed (Participants) | 4 | 6
  Day 15 | 82.9 (25.42) | 84.1 (7.70)

8. Secondary Outcome: Time to Reach Cmax (Tmax) of PEGPH20
Description: Samples were analyzed for PEGPH20 concentration using a validated electrochemiluminescence immunoassay. Plasma samples to assess the potential effects of NAB+GEM on PEGH20 PK were collected in the PAG treatment group in the run-in phases (Run-in Phase 1: Original PEGPH20 formulation [3.5 mg/mL], and Run-in Phase 2: New PEGPH20 formulation [0.3 mg/mL]).
Time Frame: Pre-PEGPH20 dosing and 15 minutes, 1 hour, 2 hours, and 4 hours post-PEGPH20 dosing on Days 1 and 15 of Cycle 1
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Run-in Phase 1-PAG: PEGPH20 (Original Formulation) + NAB + GEM | Run-in Phase 2- PAG: PEGPH20 (New Formulation) + NAB + GEM
Number analyzed (Participants) | 6 | 8
hours
  Day 1: number analyzed (Participants) | 5 | 8
  Day 1 | 0.430 [0.33 to 4.17] | 0.865 [0.33 to 4.20]
  Day 15: number analyzed (Participants) | 4 | 6
  Day 15 | 0.790 [0.00 to 1.93] | 0.810 [0.42 to 2.28]

9. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Last Quantifiable Concentration (AUC0-last) of PEGPH20
Description: as for outcome 8
Time Frame: Pre-PEGPH20 dosing and 15 minutes, 1 hour, 2 hours, and 4 hours post-PEGPH20 dosing on Days 1 and 15 of Cycle 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Run-in Phase 1-PAG: PEGPH20 (Original Formulation) + NAB + GEM | Run-in Phase 2- PAG: PEGPH20 (New Formulation) + NAB + GEM
Number analyzed (Participants) | 6 | 8
hours*ng/mL
  Day 1: number analyzed (Participants) | 5 | 7
  Day 1 | 1837.93575 (374.093974) | 2143.30319 (491.270018)
  Day 15: number analyzed (Participants) | 4 | 5
  Day 15 | 2807.94210 (687.004217) | 2423.01690 (261.783892)

ADVERSE EVENTS:
Time Frame: From first exposure to any study drug (PEGPH20, NAB, GEM) through 30 days after end of treatment visit (maximum exposure: 30.72 months for PAG and 20.27 months for AG)
Description: AEs were analyzed on safety population, which included all participants who received at least 1 dose of study drug. AE data was collected and reported combined for both phases per treatment arm (PAG and AG).
  All-cause mortality was reported for all randomized participants.
Arm/Group | PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine | AG: Nab-paclitaxel + Gemcitabine
All-Cause Mortality (participants affected / at risk) | 131/166 | 87/113
Serious Adverse Events (participants affected / at risk) | 101/160 | 58/100
Other Adverse Events (participants affected / at risk) | 157/160 | 98/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine (N=160) | AG: Nab-paclitaxel + Gemcitabine (N=100)
Sepsis (Infections and infestations) | 13 | 11
Pneumonia (Infections and infestations) | 8 | 2
Bacteraemia (Infections and infestations) | 3 | 4
Urinary tract infection (Infections and infestations) | 3 | 2
Device related infection (Infections and infestations) | 3 | 1
Liver abscess (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 1 | 2
Clostridium difficile infection (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 1
Peritonitis (Infections and infestations) | 2 | 0
Urosepsis (Infections and infestations) | 1 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 4
Vomiting (Gastrointestinal disorders) | 8 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 3 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 2
Large intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 2 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 11 | 2
Asthenia (General disorders) | 3 | 1
Fatigue (General disorders) | 3 | 1
Generalised oedema (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 1
Chills (General disorders) | 0 | 1
Extravasation (General disorders) | 1 | 0
Incarcerated hernia (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 6 | 5
Neutropenia (Blood and lymphatic system disorders) | 7 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Splenic haematoma (Blood and lymphatic system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 12 | 4
Failure to thrive (Metabolism and nutrition disorders) | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Vitamin K deficiency (Metabolism and nutrition disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 8 | 4
Atrial flutter (Cardiac disorders) | 2 | 2
Cardiac failure (Cardiac disorders) | 1 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Device occlusion (Product Issues) | 0 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Retinal vascular disorder (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
White blood cell count decreased (Investigations) | 2 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Transfusion-associated dyspnoea (Injury, poisoning and procedural complications) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 2
Mental status changes (Psychiatric disorders) | 0 | 2
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 4
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 4 | 0
Encephalopathy (Nervous system disorders) | 0 | 2
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 4 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 1 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 2
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Malignant hypertension (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PAG: PEGPH20 + Nab-paclitaxel + Gemcitabine (N=160) | AG: Nab-paclitaxel + Gemcitabine (N=100)
Anaemia (Blood and lymphatic system disorders) | 63 | 41
Leukopenia (Blood and lymphatic system disorders) | 15 | 7
Lymphopenia (Blood and lymphatic system disorders) | 8 | 5
Neutropenia (Blood and lymphatic system disorders) | 53 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 41 | 17
Sinus tachycardia (Cardiac disorders) | 6 | 5
Tachycardia (Cardiac disorders) | 15 | 7
Vision blurred (Eye disorders) | 13 | 5
Abdominal distension (Gastrointestinal disorders) | 16 | 9
Abdominal pain (Gastrointestinal disorders) | 51 | 28
Abdominal pain lower (Gastrointestinal disorders) | 9 | 3
Abdominal pain upper (Gastrointestinal disorders) | 10 | 5
Ascites (Gastrointestinal disorders) | 13 | 5
Constipation (Gastrointestinal disorders) | 58 | 36
Diarrhoea (Gastrointestinal disorders) | 81 | 49
Dry mouth (Gastrointestinal disorders) | 11 | 5
Dyspepsia (Gastrointestinal disorders) | 7 | 7
Dysphagia (Gastrointestinal disorders) | 12 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 4
Nausea (Gastrointestinal disorders) | 91 | 53
Stomatitis (Gastrointestinal disorders) | 19 | 11
Vomiting (Gastrointestinal disorders) | 51 | 33
Asthenia (General disorders) | 23 | 17
Chills (General disorders) | 23 | 9
Fatigue (General disorders) | 124 | 72
Gait disturbance (General disorders) | 10 | 5
Influenza like illness (General disorders) | 8 | 1
Mucosal inflammation (General disorders) | 12 | 5
Non-cardiac chest pain (General disorders) | 10 | 1
Oedema peripheral (General disorders) | 119 | 41
Pain (General disorders) | 8 | 5
Peripheral swelling (General disorders) | 13 | 5
Pyrexia (General disorders) | 47 | 30
Candida infection (Infections and infestations) | 16 | 5
Cellulitis (Infections and infestations) | 5 | 6
Oral candidiasis (Infections and infestations) | 14 | 4
Pneumonia (Infections and infestations) | 10 | 1
Upper respiratory tract infection (Infections and infestations) | 12 | 7
Urinary tract infection (Infections and infestations) | 22 | 11
Contusion (Injury, poisoning and procedural complications) | 10 | 3
Fall (Injury, poisoning and procedural complications) | 15 | 8
Alanine aminotransferase increased (Investigations) | 33 | 12
Aspartate aminotransferase increased (Investigations) | 26 | 12
Blood alkaline phosphatase increased (Investigations) | 14 | 11
Blood bilirubin increased (Investigations) | 14 | 1
Lymphocyte count decreased (Investigations) | 12 | 2
Neutrophil count decreased (Investigations) | 33 | 22
Platelet count decreased (Investigations) | 38 | 10
Weight decreased (Investigations) | 32 | 17
White blood cell count decreased (Investigations) | 29 | 9
Decreased appetite (Metabolism and nutrition disorders) | 75 | 39
Dehydration (Metabolism and nutrition disorders) | 30 | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 18 | 12
Hypoalbuminaemia (Metabolism and nutrition disorders) | 27 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 13 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 38 | 22
Hypomagnesaemia (Metabolism and nutrition disorders) | 19 | 13
Hyponatraemia (Metabolism and nutrition disorders) | 26 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 92 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 19 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 43 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 7
Dizziness (Nervous system disorders) | 39 | 25
Dysgeusia (Nervous system disorders) | 48 | 22
Headache (Nervous system disorders) | 13 | 14
Neuropathy peripheral (Nervous system disorders) | 50 | 32
Paraesthesia (Nervous system disorders) | 9 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 18 | 15
Syncope (Nervous system disorders) | 3 | 6
Anxiety (Psychiatric disorders) | 18 | 13
Depression (Psychiatric disorders) | 17 | 12
Insomnia (Psychiatric disorders) | 31 | 17
Dysuria (Renal and urinary disorders) | 8 | 2
Pollakiuria (Renal and urinary disorders) | 6 | 7
Urinary retention (Renal and urinary disorders) | 8 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 23
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 30 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 | 31
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 25 | 14
Hiccups (Respiratory, thoracic and mediastinal disorders) | 18 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 18 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 61 | 39
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 2
Erythema (Skin and subcutaneous tissue disorders) | 7 | 5
Night sweats (Skin and subcutaneous tissue disorders) | 7 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 8
Rash (Skin and subcutaneous tissue disorders) | 25 | 21
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15 | 7
Deep vein thrombosis (Vascular disorders) | 12 | 7
Flushing (Vascular disorders) | 10 | 0
Hypertension (Vascular disorders) | 8 | 3
Hypotension (Vascular disorders) | 35 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT01839487/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT01839487/SAP_001.pdf